CLINICAL TRIAL: NCT06890650
Title: Efficacy of Microbiome Manipulation Strategies (fecAL Microbial Transplantation OR CDED OR Both) in Combination Standard Medical Therapy for Induction and Maintenance of Remission in Mild to Moderate tReatment naÃive Active Crohns Disease (ALTER-CD): a Multicentre Double-blind Factorial Randomized Controlled Trial
Brief Title: A Study to Evaluate the Effect of Fecal Transplant and Dietary Changes on Disease Activity in Patients With Newly Diagnosed Active Crohn Disease
Acronym: ALTER-CD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Dayanand Medical College and Hospital (Other); Institute of Medical Sciences of the Banaras Hindu University, India (Other); Lokmanya Tilak Municipal Medical College and Hospital (Other); Lisie Hospital (Other); Indraprastha Institute of Information Technology Delhi (Other); Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Prof. Vineet Ahuja, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AIIMSA2989/03.01.2025; EMDR/CARE/12/2023-0000572 (Other Grant/Funding Number: Indian Council of Medical Research)
Record Dates: First submitted 2025-03-03; First posted 2025-03-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
Keywords: Randomized controlled trial; factorial design; Fecal microbiota transplantation; Crohn disease; Crohn disease exclusion diet
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fecal Microbiota Transplantation(FMT) with Crohns disease exclusion diet(CDED) (Experimental): 1. Oral vancomycin 500 mg BD for 3 days before first FMT 2. FMT via colonoscopy at 0, 2 and 6 weeks followed by (if treatment responder) 8 weekly during maintenance between 10 to 48 weeks
  Interventions: Other: Fecal Microbial Transplantation; Other: Crohns disease exclusion diet
- Fecal microbiota transplantation(FMT) and sham diet (Experimental): 1. Oral vancomycin 500 mg BD for 3 days before first FMT 2. FMT via colonoscopy at 0, 2 and 6 weeks followed by (if treatment responder) 10 weeks and then 8 weekly during maintenance between 10 to 42 weeks 3. Diet counselling for 48 weeks
  Interventions: Other: Fecal Microbial Transplantation; Other: Sham diet
- Crohns Disease Exclusion Diet(CDED) and sham transplantation (Experimental): 1. Oral placebo 1 BD for 3 days before first FMT 2. Sham transplantation (clean water) via colonoscopy at 0, 2 and 6 weeks followed by (if treatment responder) 8 weekly during maintenance between 10 to 48 weeks 3.Crohns Disease Exclusion Diet for 48 weeks
  Interventions: Other: Sham transplantation; Other: Crohns disease exclusion diet
- Sham transplantation with Sham diet (Sham Comparator): 1.Oral placebo 1 BD for 3 days before first sham transplantation 2. Sham colonoscopy with instillation of saline at 0, 2, and 6 weeks followed by (if treatment responder) - 8-weekly during maintenance between 10 to 48 weeks
  Interventions: Other: Sham transplantation; Other: Sham diet

INTERVENTIONS:
Other: Fecal Microbial Transplantation — This will involve colonoscopic instillation of fecal transplant
  Arms: Fecal Microbiota Transplantation(FMT) with Crohns disease exclusion diet(CDED); Fecal microbiota transplantation(FMT) and sham diet
Other: Sham transplantation — Sham FMT will involve saline infusion via colonoscopy
  Arms: Crohns Disease Exclusion Diet(CDED) and sham transplantation; Sham transplantation with Sham diet
Other: Crohns disease exclusion diet — The modified diet plan will be given to each study participant
  Arms: Crohns Disease Exclusion Diet(CDED) and sham transplantation; Fecal Microbiota Transplantation(FMT) with Crohns disease exclusion diet(CDED)
Other: Sham diet — Dietary counselling alone
  Arms: Fecal microbiota transplantation(FMT) and sham diet; Sham transplantation with Sham diet

SUMMARY:
Dysbiosis can be rectified by several methods: antibiotics, prebiotics, probiotics, dietary modulation, and fecal microbiota transplantation. There has been limited success with the isolated use of antibiotics and pre/probiotics in the treatment of IBD. Among the measures of dietary manipulation, the use of exclusive enteral nutrition (EEN) has shown superior, or at least equivalent, efficacy compared with steroids in pediatric CD. Although the results in adults are not as encouraging, recent cohort studies in patients with complicated CD have shown good success rates. Definite exclusion diets that exclude pro-inflammatory dietary constituents have also been tested with good clinical efficacy in patients with CD, who even failed treatment with anti-TNF agents. Various dietary approaches, inclusive of exclusive enteral nutrition, partial enteral nutrition, and Crohn's disease exclusion diet have been reported to be of benefit and are associated with changes in gut microbiome. Fecal microbiota transplantation (FMT) defined as the infusion of fecal suspension from a healthy individual into the gastrointestinal tract of an individual with GI disease carries a diverse population of microbiota and their metabolites and has been tested with varying efficacy in IBD. In general, FMT has shown good success rates in randomized control trials in patients with UC who failed conventional agents. Although limited small RCTs exist in CD, cohort studies have also shown good success rates. Therefore, the use of FMT in addition to standard medical therapy, is a concept that has not been previously explored and forms the basis for the present study. Therefore, a well-powered RCT is required to resolve the role of FMT in CD. In this study, patients will be recruited in four arms. Group A includes FMT+CDED+SMT, in Group B FMT+SMT+SHAM DIET, in Group C Sham FMT+CDED+SMT, in Group D Sham FMT+ Sham Diet+ SMT given. 168 patients will be recruited across 6 centers for around 3 years. Follow-up of the patient will be done at 0,2,6 and 10 weeks and 8 weekly up to 48 weeks.

DETAILED DESCRIPTION:
This study is a multi-center, double-blind, factorial randomized controlled trial designed to evaluate the efficacy of microbiome manipulation strategies using fecal microbiota transplantation (FMT), Crohn's Disease Exclusion Diet (CDED), or their combination in treatment-naïve patients with mild to moderate active Crohn's Disease (CD).

Study Setting

The trial is conducted at six FMT centers across India, with one additional center dedicated to microbiome analysis:

AIIMS, New Delhi, India Dayanand Medical College, Ludhiana, India PGIMER, Chandigarh, India Lisie Hospital, Kochi, India IMS, BHU, Varanasi, India Sion Hospital, Mumbai, India IIIT-Delhi, India(for microbiome analysis)

Intervention Details:

Fecal Microbiota Transplantation (FMT)- Patients receive a 3-day course of oral vancomycin (500 mg BD) before the first FMT.

Freshly prepared 50 g stool is used for each FMT, and the transplant is administered within 4 hours of preparation.

FMT is delivered via colonoscopy at weeks 0, 2, and 6, followed by 8-weekly maintenance sessions for responders at weeks 10, 18, 26, 34, 42.

Multiple donors (n≥2) are used to ensure microbiome diversity. The first FMT session is instilled in the right colon/terminal ileum post bowel preparation, whereas maintenance sessions involve left-colon infusion without bowel preparation.

Crohn's Disease Exclusion Diet (CDED)- Patients assigned to CDED follow a phased dietary protocol designed to limit exposure to pro-inflammatory dietary components and enhance gut microbiome stability.

CDED consists of an induction and maintenance phase, with structured dietary charts and counseling provided by a dietitian.

Compliance is monitored via telephonic interviews and a dedicated diet tracking app (IBD NutriCare).

Sham Interventions- Sham FMT: Patients receive sterile water or saline infusions via colonoscopy at the same time points as FMT.

Sham Diet: Patients receive general dietary advice but do not follow the CDED protocol.

Randomization and Blinding- Central randomization is conducted using a secure web-based system (REDCap), utilizing stratified randomization based on disease extent.

The study follows a double-blind approach:

Blinded: Patients, clinical assessors, and endoscopic scorers. Unblinded: Endoscopists administering FMT/sham FMT and dietitians providing dietary counseling.

Oral vancomycin and placebo capsules are identically packed to maintain blinding.

Data Collection and Assessments- Baseline Assessments (Week 0) Clinical Assessment: Crohn's Disease Activity Index (CDAI), symptom scoring, and dietary adherence evaluation.

Laboratory Tests: Hemogram, renal/liver function, CRP, ESR, fecal calprotectin, and microbiome profiling.

Endoscopy: SES-CD scoring with high-definition endoscopic video recording. Histology: Biopsy samples are analyzed using Distribution Chronicity and Activity (DCA) scoring.

Follow-up Assessments- Clinical assessments at weeks 0, 2, 4, 6, 10, and every 8 weeks thereafter. Endoscopic assessments at baseline, week 10, and week 48, with central reading of all videos.

Fecal microbiome analysis at baseline, week 10, and week 48. Safety and Monitoring- Adverse Events (AEs) graded per CTCAE criteria (Grades 1-5). Serious Adverse Events (SAEs) include hospitalization, life-threatening conditions, or death.

DSMB reviews interim safety data at week 10 and 24. Emergency unblinding is permitted for critical medical decisions. Data Management- Data is collected using REDCap, with role-based access controls. Endoscopic images and videos are securely stored for centralized analysis. Microbiome sequencing data is processed at IIIT-Delhi. Statistical Considerations- Sample size calculation: 168 patients (42 per arm, 90% power).

Analysis Plan:

Intention-to-treat (ITT) and per-protocol (PP) analyses. Longitudinal mixed-effects modeling for microbiome shift

ELIGIBILITY:
Inclusion Criteria:

1. Patients with treatment-naive Crohns disease accessible with ileocolonoscopy
2. Symptom onset of less than 12 months
3. Mild to moderate disease activity with endoscopically active disease

   1. CDAI of greater than 150 and less than 450
   2. SES-CD of or equal to or greater than 6 (or equal to or greater than 4 if isolated ileal disease)
4. Aged between 18-75 years

Exclusion Criteria:

1. Patients with severe disease (CDAI greater than 450, SES-CD greater than 16) or requiring hospitalization
2. Patients who have been received on corticosteroids, immunosuppressants (azathioprine/ 6- mercaptoprine/methotrexate) for greater than 2 weeks
3. Biologicals or small molecule exposure
4. Stricturing (non-passable stricture), fistulising phenotype or perianal fistula/abscess
5. L4 disease
6. Pregnant or lactating women
7. Previous surgery for CD
8. Declining consent
9. Not willing for FMT/Dietary advise
10. Patients with current or recent history of clinically severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurological disease.
11. Positive assay or stool culture for pathogens (ova and parasite examination, bacteria) or positive test for Clostridioides difficile toxin at screening#
12. Patients infected with human immunodeficiency virus (HIV) # The patients with positive assay will be treated appropriately and tests will be repeated. Those with negative assay and persistent activity will be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with clinical remission and endoscopic response at week 10 | 10 weeks
  Proportion of patients with clinical remission (defined as CDAI less than 150) and endoscopic response( defined decline in SES-CD by gretaer than 50%).
Proportion of patients with clinical remission and endoscopic remission at week 48 | 48 weeks
  Proportion of patients with clinical remission (defined as Crohn's disease activity index less than 150) and endoscopic remission (defined as Simple Endoscopic Score for Crohn's disease patients less than 3)

SECONDARY OUTCOMES:
Proportion of patients with clinical response at Week 10 | 10 weeks
  Proportion of patients with clinical response is defined as either CDAI decrease from baseline of at least 70 points or CDAI less than 150
Proportion of patients with PRO2 Remission at Week 10 | 10 weeks
  Proportion of patients with PRO2 Remission which is defined as Abdominal pain subscore of not more than 1 (on a scale of 0-3) and liquid or very soft stool (Bristol stool scale type 6 or 7) frequency subscore of not more than 3 calculated as a mean of 7 day count
Proportion of patients with endoscopic response at Week 10 | 10 weeks
  Proportion of patients with endoscopic response which is defined as 50% reduction from baseline on SES-CD
Fecal microbiome and metabolite signature between responders and non-responders at week 10 | 10 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Proportion of patients with biomarker remission at Week 10 | 10 weeks
  Proportion of patients with biomarker remission which is defined as fecal calprotectin ≤150 mcg/g
Proportion of patients with adverse events at Week 10 | 10 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))
Proportion of patients with clinical response at Week 48 | 48 weeks
  Proportion of patients with clinical response is defined as either CDAI decrease from baseline of at least 70 points or CDAI less than 150
Proportion of patients with PRO2 remission at Week 48 | 48 weeks
  Proportion of patients with PRO2 remission is defined as Abdominal pain subscore of not more than 1 (on a scale of 0-3) and liquid or very soft stool (Bristol stool scale type 6 or 7) frequency subscore of not more than 3 calculated as a mean of 7 day count
Proportion of patients with endoscopic response at Week 48 | 48 weeks
  Proportion of patients with endoscopic response defined as 50% reduction from baseline on SES-CD
Proportion of patients with Endoscopic remission at Week 48 weeks | 48 weeks
  Proportion of patients with Endoscopic remission defined as a SES-CD score of 2 or less
Proportion of patients with corticosteroid-free clinical remission at Week 48 | 48 weeks
  Proportion of patients with corticosteroid-free clinical remission is defined as the CDAI<150 with no exposure to steroids over the previous 8 weeks
Fecal microbiome and metabolite signature between responders and non-responders at Week 48 | 48 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Proportion of patients with biomarker remission at Week 48 | 48 weeks
  Proportion of patients with biomarker remission which is defined as fecal calprotectin ≤150 mcg/g
Proportion of patients with adverse event at Week 48 | 48 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))
Proportion of patients with adverse event at Week 6 | 6 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))
Proportion of Patients Experiencing Adverse Events at Week 26 | 26 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))

CONTACTS AND LOCATIONS:
Overall Officials: Prof Vineet Ahuja, DM Gastroenterology, Principal Investigator — Department of Gastroenterology, AIIMS, New Delhi
Locations (6):
- India (6):
  - Department of Gastroenterology, Lisie Hospital, Kochi, Kerala
  - Lokmanya Tilak Municipal General Hospital and Lokmanya Tilak Municipal Medical College, Sion, Mumbai, Maharashtra
  - Department of Gastroenterology and Human Nutrition, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Department of Gastroenterology, Dayanand Medical College, Ludhiana, Punjab
  - Department of Gastroentrology, Postgraduate Institute of Medical Education and Research, Chandigarh, Punjab/Haryana
  - Department of Gastroenterology, Institute of Medical Sciences, Banaras Hindu University, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No